CLINICAL TRIAL: NCT02727569
Title: Quantification of Agreement and Variability Characteristics of a Newly Developed Visual Field Algorithm With the Reference Standard: an Observational Study
Brief Title: Quantification of Agreement and Variability of a Newly Developed Visual Field Algorithm With the Reference Standard
Acronym: vFAST
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GART1046
Record Dates: First submitted 2016-03-15; First posted 2016-04-04 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Glaucoma; Healthy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Feasibility Study: 10 subjects. Subjects will performed two different versions of the new visual field algorithm with DLS (differential light sensitivity) strategies. Two repeats of each strategy will be performed.
  Interventions: Device: New visual field algorithm with DLS
- Clinical evaluation study: 100 subjects. Subjects will performed a visual field assessment with the new visual field algorithm with MMDT (Moorfields Motion Displacement Test) and DLS -like stimuli and a commercial available SITA algorithm (DLS-like strategy). Two repeats of each strategy will be performed.
  Interventions: Device: New visual field algorithm with DLS; Device: SITA algorithm; Device: New visual field algorithm with MMDT

INTERVENTIONS:
Device: New visual field algorithm with DLS — Mathematical model (software based) to derive retinal sensitivity.
Device: SITA algorithm — Mathematical model (software based) to derive retinal sensitivity. Commercially available.
  Groups: Clinical evaluation study
Device: New visual field algorithm with MMDT — Mathematical model (software based) to derive retinal sensitivity.
  Groups: Clinical evaluation study

SUMMARY:
This study aims to compare two types of visual field test; retinal sensitivity values obtained with the reference standard Swedish Interactive Thresholding Algorithm (SITA) of the standard visual field test and with a newly developed test algorithm. The new test is a visual field test presented on a flat-panel monitor and has two modes: differential light sensitivity (DLS; equivalent to the standard visual field test) and the Moorfields Motion Displacement Test (MMDT). DLS sensitivity and DLS measurement variability will be determined and compared between the SITA algorithm of the standard visual field test and the new visual field test on the flat-panel monitor. The measurement variability of the MMDT will be quantified.

The long-term goal is to reduce test variability below that observed in SITA by 20%, whilst producing comparable measurements (contrast threshold values) for comparable test duration.

DETAILED DESCRIPTION:
Standard Automated Perimetry (SAP) is currently the standard test for screening and monitoring visual loss owing to glaucoma. This test requires the patient to sit at a machine, looking at a central light and pressing a button whenever small spots of light appear in the peripheral vision. Traditionally these spots of light are projected into a bowl (concave surface), but more recently, computer monitors have been used. Other techniques are also now available such as the Moorfields Motion Displacement Test, where patients are required to press a button each time they see a vertical line on the screen wiggle. This test has been shown to have advantages over SAP, namely, to be tolerant to the effects of cataract and refractive error.

In clinical settings, the Humphrey Visual Field Analyzer (Zeiss Meditec) is the most used visual field test in the UK. It employs a SAP strategy coupled with the Swedish Interactive Thresholding Algorithm (SITA), which is used to derive retinal sensitivity. Visual field measurements are very variable, requiring many tests over a long period to determine the extent of vision loss. In addition to the inconvenience caused to patients, the contribution of these many tests to the financial burden on the NHS is increasing with the growing aging population. As glaucoma is a chronic disease, patients need lifelong monitoring, requiring multiple tests and clinic visits. To address these unmet needs, the investigators have developed a new algorithm that can be used to monitor glaucoma.

The investigators wish to carry out a study, which will allow them to compare agreement between SITA and a newly developed test algorithm. Measurement variability will be determined and compared between strategies. The long-term goal is to reduce test variability and the test time observed in SITA, whilst producing comparable contrast threshold values.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity of 6/12 or better in the test eye
* No ocular morbidity other than glaucoma; early lens opacity and prior cataract surgery are acceptable

Healthy eyes

* Central 30° visual field within normal limits on the 24-2 test (MD within 95 % CI and glaucoma hemifield test within normal limits).

Glaucoma eyes

* More than two reliable visual fields with reproducible defects
* IOP < 30 mmHg

Exclusion Criteria:

* Any systemic disease which is likely to affect visual performance in a short period of time
* Inability to steadily fixate on the test (e.g. individuals who have nystagmus or macular degeneration)
* Eyes with unreliable visual fields (defined as false positive responses >15%)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited using three methods:
  1. The volunteer database of the Glaucoma Research Unit. Letters will be sent to patients/healthy controls, who in the past agreed to be contacted for research purposes. Written information about the project will be sent with the letters.
  2. Records screening. Patients' records will be screened in advance or during their clinical appointment. Persons identified as meeting the inclusion criteria will be invited to join the study, whereupon written information about the project will be given to the patient. Patients will be invited to join the study by letter, prior to their clinical appointment or in person on the day of the appointment.
  3. Invitation of accompanying persons and staff. It is anticipated that spouses and acquaintances of existing subjects, as well as staff at the research site, Moorfields Eye Hospital and UCL Institute of Ophthalmology, may offer their participation as healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
To quantify the threshold difference in the test-retest variability of DLS obtained with the new algorithm and the SITA algorithm. To quantify the threshold test-retest variability of the MMDT with the new algorithm. | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
To quantify the difference in DLS thresholds measured with the new and SITA algorithms across all retinal locations and for a range of visual field sensitivities. | Through study completion, an average of 1 year.
To determine whether any differences in thresholds obtained on the two algorithms vary with retinal eccentricity and stimulus energy. Mean difference for each location will be reported in decibels. | Through study completion, an average of 1 year.
To determine whether any differences in test-retest variability obtained on the two algorithms vary with retinal eccentricity and stimulus energy. Mean difference between test-retest for each location will be reported in decibels. | Through study completion, an average of 1 year.
Participants preference for a more reliable visual fields test or for having a shorter test (questionnaire). | Through study completion, an average of 1 year.
Participants preference of test strategy, MMDT or DLS (questionnaire). | Through study completion, an average of 1 year.
Participants preference of test algorithm, newly developed algorithms or the SITA algorithm (questionnaire). | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: David Garway-Heath, MD, Principal Investigator — NIHR Biomedical Research Centre, Moorfields Eye Hospital and UCL Institute of Ophthalmology
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom